CLINICAL TRIAL: NCT02220244
Title: Effect of MD1003 in Chronic Visual Loss Related to Optic Neuritis in Multiple Sclerosis: a Pivotal Randomized Double Masked Placebo Controlled Study
Brief Title: Effect of MD1003 in Chronic Visual Loss Related to Optic Neuritis in Multiple Sclerosis
Acronym: MS-ON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD1003CT2013-01MS-ON; 2013-002112-27 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis (MS); optic neuritis; visual defect; visual loss; relapsing remitting multiple sclerosis (RRMS); primary progressive multiple sclerosis (PPMS); secondary progressive multiple sclerosis (SPMS)
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; Vision Disorders; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MD1003 (Experimental): MD1003 100mg capsule, 1 capsule TID for 12 months
  Interventions: Drug: MD1003 100mg capsule
- Placebo (Placebo Comparator): Placebo capsule, 1 capsule TID for 6 months, then switch to MD1003 100mg capsule, 1 capsule TID for 6 months
  Interventions: Drug: MD1003 100mg capsule

INTERVENTIONS:
Drug: MD1003 100mg capsule

SUMMARY:
The purpose of this study is to demonstrate the superiority of MD1003 over placebo in the visual improvement of patients suffering from chronic visual loss resulting from multiple sclerosis related optic neuritis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis criteria of MS fulfilling revised Mc Donald criteria (2010)
2. Uni-or bilateral optic neuropathy with worst eye VA≤ 5/10 confirmed at 6 months
3. Worsening of visual acuity during the last three years
4. Informed consent prior to any study procedure
5. Patient aged 18-75 years

Exclusion Criteria:

1. Optic neuritis relapse within the three months before inclusion
2. Normal RNFL at OCT
3. Presence of other ocular pathology (glaucoma, cataract, retinopathy, anterior uveitis, myopia>7 dioptrics, intraocular pressure>20 mm Hg, amblyopia, retinal or optic head abnormalities (drusen, tilted disc)
4. Bilateral visual acuity <1/20
5. Visual impairment caused by ocular flutter or nystagmus
6. Pregnancy or childbearing potential woman without contraception
7. Any general chronic handicapping disease other than MS
8. New treatment introduced less than 3 months prior to inclusion or less than 1 month for Fampridine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the best corrected visual acuity at 100% contrast | Baseline, 6 months
  Best corrected visual acuity using the ETDRS logMar chart at 100% contrast

SECONDARY OUTCOMES:
Visual field mean deviation change from baseline | Baseline, 6 months, 12 months
  Visual field analyses are performed using the standard automated perimetry method
Reappearance or improvement of the P00 wave on Visual Evoked Potential | Baseline, 6 months, 12 months
  Two parameters will be evaluated: (1) presence of a clear P100 wave, (2) P100 latency
Optical Coherence Tomography | Baseline, 6 months, 12 months
  Values of RNFL thickness and macular volume

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Tourbah, MD, PhD, Principal Investigator — Hopital Maison Blanche; Frederic Sedel, MD, PhD, Study Director — MedDay Pharmaceuticals SA
Locations (20):
- France (19):
  - Hopital Pellegrin, Bordeaux
  - Hopital de la cote de Nacre, Caen
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital general du Bocage, Dijon
  - CHRU de Lille, Lille
  - Hopital Pierre Wertheimer, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - Hopital Central, Nancy
  - Hopital Nord Laennec, Nantes
  - Hopital Pasteur, Nice
  - Centre hospitalier national d'ophtalmologie des Quinze Vingts, Paris
  - Groupe hospitalier la Pitie-Salpetriere, Paris
  - Fondation Rothschild, Paris
  - Centre hospitalier Intercommunal Poissy/Saint-Germain-en-Laye, Poissy
  - Hopital Maison Blanche, Reims
  - Hopital Pontchaillou, Rennes
  - Hopital de Hautepierre, Strasbourg
  - Hopital Purpan, Toulouse
- UCL Institute of Neurology, London, United Kingdom

REFERENCES:
- [Derived] Tourbah A, Gout O, Vighetto A, Deburghgraeve V, Pelletier J, Papeix C, Lebrun-Frenay C, Labauge P, Brassat D, Toosy A, Laplaud DA, Outteryck O, Moreau T, Debouverie M, Clavelou P, Heinzlef O, De Seze J, Defer G, Sedel F, Arndt C. MD1003 (High-Dose Pharmaceutical-Grade Biotin) for the Treatment of Chronic Visual Loss Related to Optic Neuritis in Multiple Sclerosis: A Randomized, Double-Blind, Placebo-Controlled Study. CNS Drugs. 2018 Jul;32(7):661-672. doi: 10.1007/s40263-018-0528-2. PMID 29808469